CLINICAL TRIAL: NCT01645774
Title: Comparing Pain and Bruising of Subcutaneous Heparin Injection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tayebe Pourghaznein, faculty member,MSc of Nursing, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: interventional
Record Dates: First submitted 2012-05-19; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-06

CONDITIONS: Pain; Bruising
Keywords: subcutaneous injection heparin; injection duration; bruising pain; decrease pain; decrease bruising
MeSH Terms: conditions — Pain; Contusions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10s injections duration (Experimental): 10s injections duration
  Interventions: Procedure: 10s injections duration
- 10s injection duration , waiting 10s (Experimental): 10s injection duration and waiting 10s before withdrawing the needle
  Interventions: Procedure: 10s injection duration and waiting 10s before withdrawing the needle
- 15s injection duration,waiting 5s (Experimental): 15s injection duration and waiting 5s before withdrawing the needle
  Interventions: Procedure: 15s injection duration and waiting 5s before withdrawing the needle
- 5s injection duration , waiting 15s (Experimental): 5s injection duration and waiting 15s before withdrawing the needle
  Interventions: Procedure: 5s injection duration and waiting 15s before withdrawing the needle

INTERVENTIONS:
Procedure: 10s injections duration — 10s injections duration
  Arms: 10s injections duration
Procedure: 10s injection duration and waiting 10s before withdrawing the needle — 10s injection duration and waiting 10s before withdrawing the needle
  Arms: 10s injection duration , waiting 10s
Procedure: 15s injection duration and waiting 5s before withdrawing the needle — 15s injection duration and waiting 5s before withdrawing the needle
  Arms: 15s injection duration,waiting 5s
Procedure: 5s injection duration and waiting 15s before withdrawing the needle — 5s injection duration and waiting 15s before withdrawing the needle
  Arms: 5s injection duration , waiting 15s

SUMMARY:
Subcutaneous heparin injection is one of the most frequent nurses' clinical care. This study aimed to Identify and compare the effects of four different injection duration on pain and bruising associated with subcutaneous injection of heparin in 90 patients. Four injection methods were used for them:

A: 10s injections duration

B: 10s injection duration and waiting 10s before withdrawing the needle

C: 15s injection duration and waiting 5s before withdrawing the needle

D: 5s injection duration and waiting 15s before withdrawing the needle.

Bruising was measured by a flexible millimeter ruler 48h after each injection; and pain was measured by pain visual analogue scale immediately after the injection. Data will be analyzed by SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Inclination to participate in the study; filling out the form of conscious satisfaction
* Ability to answer the questions and determining the rate of pain
* Not being affected by blood clotting difficulties, tissue damages, injuries, and bruises in the site of injection.

Exclusion Criteria:

* Death,
* Discharge

Ages: 53 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
decrease pain | up to 6 months
  pain was measured by pain visual analogue scale immediately after the injection.
bruising | up to 6 months
  Bruising was measured by a flexible millimeter ruler 48h after each injection